CLINICAL TRIAL: NCT07281144
Title: Effect of Virtual Reality on Cannulation-Related Procedural Pain, Distress and Comfort Level in Hemodialysis Patients: A Randomized Controlled Study
Brief Title: Effect of Virtual Reality on Cannulation-Related Procedural Pain, Distress and Comfort Level in Hemodialysis Patients
Acronym: Hemodialysis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, ezgi mutluay yayla, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/106
Record Dates: First submitted 2025-11-26; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hemodialysis, Virtual Reality
Keywords: Arteriovenous fistula; Cannulation; Distress; Hemodialysis; Procedural pain; Virtual reality
MeSH Terms: conditions — Arteriovenous Fistula; Pain, Procedural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The routine cannulation procedure was applied to the patients in the control group. Apart from this, no additional intervention was implemented. Each patient's pain was evaluated and recorded by a nurse independent of the study during the procedure (1st measurements) with VAS and after the procedure (2st measurements). Similarly, the patient's distress was evaluated with Distress Thermometer and recorded before (1st measurements) and after the procedure (2st measurements) by a nurse independent of the study. HDCS of the patients were evaluated and recorded and immediately after the procedure was completed.
- Virtual Reality (Experimental): The intervention utilized VR-SHINECON and headsets, which were cleaned with alcohol-based disinfectant wipes before use for each patient. Patients in the intervention group were offered a choice of various nature, forest, and seaside walk videos with thematic music. The VR intervention commenced approximately three minutes before the cannulation procedure and continued until the procedure was complete. During the procedure, the patient's pain was evaluated and recorded by an independent nurse (referred to as the 1st measurement).Immediately after the procedure was completed, the patient removed the VR glasses. The Visual analogue scale, DT and Hemodialysis Comfort Scale were then assessed and recorded by the independent nurse (referred to as the 2nd measurements).
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — The intervention utilized VR-SHINECON and headsets, which were cleaned with alcohol-based disinfectant wipes before use for each patient (Figure 1). Patients in the intervention group were offered a choice of various nature, forest, and seaside walk videos with thematic music. The VR intervention commenced approximately three minutes before the cannulation procedure (immediately following the baseline assessment) and continued until the procedure was complete (approx. 5-10 minutes).
  Arms: Virtual Reality

SUMMARY:
This study aimed to determine the effects of virtual reality on procedural pain, distress and comfort levels during cannulation in hemodialysis patients.

DETAILED DESCRIPTION:
Background Virtual reality is a non-pharmacological method that reduces pain and distress and increases comfort by diverting a patient's attention. This allows individuals to gain self-control and relax during medical procedures.

Purpose: This study aimed to determine the effects of virtual reality on procedural pain, distress and comfort levels during cannulation in hemodialysis patients.

Methods: This randomized controlled study included a total of 52 patients, who were randomly assigned to either the intervention group (n=26) or the control group (n=26). Patients in the intervention group received virtual reality glasses during the procedure in addition to standard routine care, while the control group received standard routine care only. Data were collected using a Descriptive Information Form, the Visual Analogue Scale (VAS), the Distress Thermometer (DT), and the Hemodialysis Comfort Scale. Statistical analysis was performed with the level of significance set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years and older
* who had been receiving hemodialysis treatment via AVF for four-hour sessions three times per week for at least six months
* had a pain score of 0 according to the VAS before the procedure
* were not using any psychiatric medicatio
* voluntarily agreed to participate in the study

Exclusion Criteria:

* Patients were excluded if they had a diagnosed mental health disability,
* language barriers
* were using analgesic drugs within eight hours prior to the hemodialysis session
* a history of epilepsy, vertigo, anxiety, active nausea, vomiting, or headaches
* regular use of painkillers
* chronic pain disorders
* previous experience with virtual reality.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
The data were collected by the researcher by using "Descriptive Information Form" | The descriptive information form was completed in the patient's room 15-20 minutes before the cannulation procedure.
  Descriptive information form This form prepared by the researchers after reviewing relevant literature (18,21), this semi-structured form includes 12 questions focusing on the socio-demographic and medical information of the participants.
Visual Analogue Scale | During the procedure, the patient's pain was evaluated and recorded by an independent nurse (referred to as the 1st measurement). Immediately after the procedure was completed, after an average of 1-2 minutes (VAS were then assessed (2st measurement).
  This scale (VAS), originally developed by Price et al.22 and validated in Turkish for postoperative pain assessment by Eti Aslan 23, was used to quantify pain intensity. The scale consists of a 10-cm horizontal line anchored by the descriptors "no pain" and "worst imaginable pain". Participants marked their perceived pain level on the line, and the score was recorded in centimeters. Written permission for the Turkish version was secured from Eti Aslan. All VAS measurements were recorded by an independent nurse who was not involved in the intervention.
Distress Thermometer | Before the Procedure and baseline, after the procedure was completed an average of 5-10 minutes(2st measurement)
  The Distress Thermometer was first developed by Roth and colleagues for use in identifying non-pathological distress in patients undergoing cancer treatment after answering the necessary questions. The distress level is rated from 0 to 10. The practitioner expresses the distress experienced using the numbers on the thermometer. A score of zero indicates no distress, while a score of 10 indicates the highest level of distress. The green zone encompasses scores from 0 to 3. Individuals experiencing distress within this range are capable of managing their distress. The yellow zone encompasses scores from 4 to 6. A distress score in this range indicates that the individual is unable to manage their distress and requires intervention to return them to the green zone. The red zone encompasses scores from 7 to 10. Individuals experiencing distress within this range require urgent and comprehensive intervention.
Hemodialysis Comfort Scale | after the procedure was completed an average of 5-10 minutes
  This scale developed by Şahin Orak et al., is a reliable, nine-item, five-point Likert-type instrument used to assess comfort in patients receiving hemodialysis for at least six months.29 It consists of two subscales: 'Relaxation' and 'Coping.' Items are scored from 1 to 5 with Item 4 being reverse-scored. Total scores range from 9.00 to 45.00, where higher scores indicate greater comfort. Subscale ranges are 3.00-15.00 for Relaxation and 7.00-30.00 for Coping. The scale demonstrated strong reliability, with a Cronbach's alpha of 0.87 in the original Turkish validation study, and 0.80 in the present study.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - School, Mersin, Health Sciences Faculty , Tarsus University, Mersin, Turkey
  - Tarsus U, Tarsus

IPD SHARING:
Plan to Share IPD: No